CLINICAL TRIAL: NCT06273826
Title: The Implementation of the Mobile Application "Colorectal Leakage App", Based on the Dutch Leakage Score, for Early Detection of Anastomotic Leakage After Colorectal Surgeries
Brief Title: "Colorectal Leakage App" for Early Detection of Anastomotic Leakage After Colorectal Surgeries
Status: Recruiting | Type: Observational
Sponsor: National Research Oncology and Transplantology Center, Kazakhstan (Other)
Responsible Party: Principal Investigator, Meiram Mamlin, MD, Head of the colorectal division., National Research Oncology and Transplantology Center, Kazakhstan
Other Study IDs: 01
Record Dates: First submitted 2024-02-15; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Anastomotic Leak Large Intestine; Anastomotic Leak Rectum
Keywords: Anastomotic Leak; Colorectal surgery; Mobile application; Dutch Leakage Score
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal Leakage App group: This group comprises patients who will be monitored using the "Colorectal Leakage App" based on the Dutch leakage score for early detection of anastomotic insufficiency after colorectal surgeries.
  Interventions: Diagnostic Test: "Colorectal Leakage App"

INTERVENTIONS:
Diagnostic Test: "Colorectal Leakage App" — The "Colorectal Leakage App" is a mobile application designed to aid in the early detection of anastomotic insufficiency after colorectal surgeries. The app is based on the Dutch Leakage Score (DLS) algorithm, which is a standardized protocol for postoperative monitoring.

SUMMARY:
The aim of this prospective observational study is to evaluate the effectiveness of the mobile application "Colorectal Leakage App" in the early diagnosis of anastomotic leakage after colorectal surgeries at the National Research Oncology Center in Astana, Kazakhstan.

Main Questions:

1. Development, validation, and implementation of the mobile application "Colorectal Leakage App," based on the Dutch Leakage Score.
2. Evaluate the diagnostic effectiveness of the application in detecting anastomotic leakage after colorectal surgeries.
3. Determine the frequency of anastomotic leakage after colorectal surgeries performed in the colorectal surgery sector of the National Research Oncology Center in the Astana city.

Participants in the study, individuals aged 18 and above undergoing colorectal surgeries, will be monitored by the mobile application "Colorectal Leakage App" in the postoperative period for early identification of anastomotic leakage.

DETAILED DESCRIPTION:
Colorectal cancer ranks third among oncological diseases in Kazakhstan, both in men and women. Anastomotic leakage (AL) following colorectal surgeries is one of the most serious complications arising from colorectal surgical interventions. This condition is characterized by increased mortality and significant deterioration in the quality of life of patients. Additionally, the presence of AL after anterior resections for rectal cancer is associated with an increased risk of local disease recurrence. The frequency of AL varies between 2 and 19%, depending on risk factors, AL definition, and the level of anastomosis. Given the high likelihood and severe consequences of AL, a relevant task is its early detection and effective treatment.

Clinical signs of AL traditionally include fever, tachycardia, pain syndrome, purulent or fecal discharge through drainage, and dynamic bowel obstruction. These signs, combined with other clinical data, are integrated into a diagnostic-specific indicator known as the Dutch Leakage Score (DLS). This indicator is used as a standardized postoperative monitoring protocol for patients suspected of having AL, aiming to minimize delays in detecting this complication and, consequently, reduce early postoperative mortality.

In this prospective observational study, we aim to assess the effectiveness of the mobile application "Colorectal Leakage App" in the early detection of anastomotic leakage (AL) after colorectal surgeries. The study will be conducted at the National Research Oncology Center (NROC) in Astana, Kazakhstan, over one year. The primary goal is to evaluate the diagnostic effectiveness of the application in detecting AL after colorectal surgeries.

It is important to note that there is currently no up-to-date data on the number of colorectal cancer surgeries performed, and information on the frequency of AL after colorectal surgeries in the population of Kazakhstan is also lacking. Previous studies have shown that the effectiveness of the DLS algorithm is directly proportional to the frequency of AL. Therefore, it is assumed that the application of DLS may demonstrate different results in the conditions of Kazakhstan, which we also plan to measure through the "Colorectal Leakage App" mobile application.

1. Design of the study:

   Prospective observational study, where the "Colorectal Leakage App" mobile application will be implemented in daily postoperative monitoring. Additionally, an assessment of the diagnostic effectiveness of this application will be conducted.
2. Instruments and equipment:

The "Colorectal Leakage App" is a mobile application that, based on an algorithm, provides an assessment of the risk of Anastomotic Leakage (AL) in patients after colorectal surgeries. The algorithm is built on the standardized postoperative monitoring protocol called "Dutch Leakage Score". After calculating the scores, the application provides recommendations for further actions.

Primary endpoints:

1. Sensitivity, Specificity, Positive Predictive Value, Negative Predictive Value.
2. Frequency of AL after colorectal surgeries

Secondary endpoints:

1. Mortality within 30 days:.
2. Delay in the diagnosis of AL (number of days from the onset of the first signs of a leakage to the diagnosis of AL)
3. Duration of hospital stay.
4. Number of days in the ICU.
5. Number of days between surgery and detection of AL.

Postoperative monitoring with the "Colorectal Leakage App":

It is planned to implement standardized postoperative monitoring for patients who have undergone colorectal surgeries using the "Colorectal Leakage App." The application will include an algorithm based on the Dutch Leakage Score indicator. Each postoperative day, data entry at the patient's bedside will be carried out in the application.

1. Fever
2. Heart rate
3. Respiratory rate
4. Urinary production
5. Mental status
6. Clinical condition
7. Signs of ileus
8. Gastric retention
9. Fascial dehiscence
10. Abdominal pain, other than
11. wound pain
12. Increased leukocyte count, C-reactive protein (CRP), creatinine, and urea.
13. Nutritional status Based on the data analysis, the algorithm will provide recommendations regarding the necessity of conducting a computer tomography with rectal contrast.

The following information will also be collected: Preoperative risk factors for AL(age, gender, obesity, nutritional status, diabetes, cardiovascular diseases, renal insufficiency, inflammatory bowel diseases, ASAscore, bowel preparation); Surgery data (access, surgery type, anastomosis technique, duration of surgery, blood loss volume, formation of a preventive stoma, intraoperative and postoperative complications, pTNM).

Key points determining the conclusion of a patient's participation in the study will be: the detection of AL, patient discharge from the hospital, or patient death.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled patients with benign and malignant colorectal diseases undergoing surgical treatment, including the creation of anastomoses (ileocolic, colocolic, colorectal anastomoses), with or without a preventive stoma.
2. Male and female patients aged 18 years and older.
3. ECOG = 0-2; 6. Satisfactory hematological indicators and parameters of liver and kidney function.

Exclusion Criteria:

1. Participants under 18 years old.
2. Pregnant, lactating, or planning pregnancy participants.
3. ECOG>2;
4. Unresctable tumors.
5. Patient's refusal to continue participating in the study..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Scheduled patients with benign and malignant colorectal diseases undergoing surgical treatment, including the creation of anastomoses (ileocolic, colocolic, colorectal anastomoses), with or without a preventive stoma.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Diagnostic effectiveness of "Colorectal Leakage App". | 1 year
  Measurement of sensitivity, specificity, positive predictive value and negative predictive value of the mobile application "Colorectal Leakage App".
Frequency of anastomotic leakage after colorectal surgeries. | 1 year
  Measurement of frequency of anastomotic leakage after colorectal surgeries at the National Research Oncology Center (NROC) in Astana, Kazakhstan.

SECONDARY OUTCOMES:
Mortality within 30 days | 1 year
  Mortality within 30 days
Delay in the diagnosis of anastomotic leakage | 1 year
  Number of days from the onset of the first signs of a leakage to the diagnosis of anastomotic leakage..
Duration of hospital stay. | 1 year
  Duration of hospital stay.
Number of days in the ICU. | 1 year
  Number of days in the ICU.
Number of days between surgery and detection of AL. | 1 year
  Number of days between surgery and detection of AL.

CONTACTS AND LOCATIONS:
Overall Officials: Meiram Mamlin, MD, Principal Investigator — National Research Oncology Center
Locations (1):
- National Research Oncology Center, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jutesten H, Buchwald PL, Angenete E, Rutegard M, Lydrup ML. High Risk of Low Anterior Resection Syndrome in Long-term Follow-up After Anastomotic Leakage in Anterior Resection for Rectal Cancer. Dis Colon Rectum. 2022 Oct 1;65(10):1264-1273. doi: 10.1097/DCR.0000000000002334. Epub 2021 Dec 15. PMID 35482994
- [Result] Mirnezami A, Mirnezami R, Chandrakumaran K, Sasapu K, Sagar P, Finan P. Increased local recurrence and reduced survival from colorectal cancer following anastomotic leak: systematic review and meta-analysis. Ann Surg. 2011 May;253(5):890-9. doi: 10.1097/SLA.0b013e3182128929. PMID 21394013
- [Result] Akasu T, Takawa M, Yamamoto S, Yamaguchi T, Fujita S, Moriya Y. Risk factors for anastomotic leakage following intersphincteric resection for very low rectal adenocarcinoma. J Gastrointest Surg. 2010 Jan;14(1):104-11. doi: 10.1007/s11605-009-1067-4. Epub 2009 Oct 20. PMID 19841989
- [Result] Thornton M, Joshi H, Vimalachandran C, Heath R, Carter P, Gur U, Rooney P. Management and outcome of colorectal anastomotic leaks. Int J Colorectal Dis. 2011 Mar;26(3):313-20. doi: 10.1007/s00384-010-1094-3. Epub 2010 Nov 25. PMID 21107847
- [Result] Kang CY, Halabi WJ, Chaudhry OO, Nguyen V, Pigazzi A, Carmichael JC, Mills S, Stamos MJ. Risk factors for anastomotic leakage after anterior resection for rectal cancer. JAMA Surg. 2013 Jan;148(1):65-71. doi: 10.1001/2013.jamasurg.2. PMID 22986932
- [Result] Boccola MA, Lin J, Rozen WM, Ho YH. Reducing anastomotic leakage in oncologic colorectal surgery: an evidence-based review. Anticancer Res. 2010 Feb;30(2):601-7. PMID 20332477
- [Result] Kingham TP, Pachter HL. Colonic anastomotic leak: risk factors, diagnosis, and treatment. J Am Coll Surg. 2009 Feb;208(2):269-78. doi: 10.1016/j.jamcollsurg.2008.10.015. Epub 2008 Dec 4. No abstract available. PMID 19228539
- [Result] den Dulk M, Noter SL, Hendriks ER, Brouwers MA, van der Vlies CH, Oostenbroek RJ, Menon AG, Steup WH, van de Velde CJ. Improved diagnosis and treatment of anastomotic leakage after colorectal surgery. Eur J Surg Oncol. 2009 Apr;35(4):420-6. doi: 10.1016/j.ejso.2008.04.009. Epub 2008 Jun 27. PMID 18585889